CLINICAL TRIAL: NCT02359604
Title: The Gastrointestinal Microbiome of Infants With GERD and PPI Therapy: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Castellani Christoph, MD, PD Dr. med., Medical University of Graz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MUG-KCH-1
Record Dates: First submitted 2014-10-31; First posted 2015-02-10 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Gastroesophageal Reflux
Keywords: infant; ppi; proton pump inhibitor; microbiome; Microbiota
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Intervention Model Description: Longitudinal study
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Study -microbiome (Other): This is a single-arm study. The patients will serve as their own controls. The PPI administered for PPI-therapy is already FDA approved. A stool sample will be obtained for intestinal microbiome testing before PPI, under PPI and after PPI therapy.
  Interventions: Drug: PPI therapy; Procedure: Stool sample

INTERVENTIONS:
Drug: PPI therapy — PPI therapy (medication has FDA approval) for 8 weeks in children with proven GERD.
  The medication used (esomeprazole) in this trial is approved by the FDA
  Other Names: esomeprazole
Procedure: Stool sample — Stool sample will be obtained before initiation of PPI (before PPI therapy)
Procedure: Stool sample — Stool sample will be obtained 4 weeks after initiation of PPI (under PPI therapy)
Procedure: Stool sample — Stool sample will be obtained 8 weeks after termination of PPI therapy (after PPI therapy).

SUMMARY:
Proton Pump Inhibitors (PPI) are standard in the therapy of pediatric GERD. In the past it has been hypothesized, that either direct inhibition of bacterial ATPase or elevation of the pH may lead to changes in the intestinal microbiome. Small series published in adults suggest a predominance of streptococci, a possible reason for increased incidences of pneumonia under PPI therapy. Studies in children are yet scarce.

This study will include 20 infants. GERD will be verified by 24h-intraluminal impedance monitoring. All patients will have undergone conservative measures prior to initiation of PPI therapy (due to persisting symptoms). Children will receive a commercial PPI for 8 weeks (esomeprazole 1mg/kg/day). Stool samples will be collected before initiation of PPI, under PPI (4 weeks after initiation) and 8 weeks after discontinuing PPI therapy. The intestinal microbiome will be determined by 16S rDNA-based microbial community profiling by high-throughput pyrosequencing.

Data will be compared by dependent non parametric test (Wilcoxon). P-values <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

symptomatic GERD (proved by impedance monitoring) despite conservative treatment requiring PPI therapy

Exclusion Criteria:

neurological impairments

Ages: 3 Months to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2017-02-07 (Actual); Study Completion 2017-02-07 (Actual)

PRIMARY OUTCOMES:
microbial community profiling of stool to include: rate [or prevalence] of specific phyla [i.e. Proteobacteria and Firmicutes], contributing to fecal microbial communities | 16 weeks
  The change of intestinal microbiota under PPI therapy will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Castellani, MD, Principal Investigator — Dept. of Pediatric and Adolescent Surgery, Medical University Graz
Locations (1):
- Department of Pediatric and Adolescent Surgery, Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Castellani C, Singer G, Kashofer K, Huber-Zeyringer A, Flucher C, Kaiser M, Till H. The Influence of Proton Pump Inhibitors on the Fecal Microbiome of Infants with Gastroesophageal Reflux-A Prospective Longitudinal Interventional Study. Front Cell Infect Microbiol. 2017 Oct 11;7:444. doi: 10.3389/fcimb.2017.00444. eCollection 2017. PMID 29075620